CLINICAL TRIAL: NCT01322087
Title: Does the Access to Small Delicious Dishes, 24 Hours a Day, Have a Positive Effect on Nutritional Intake in Patients at Nutritional Risk?
Brief Title: Does the Access to Small Delicious Dishes, Have a Positive Effect on Nutritional Intake in Patients at Nutritional Risk?
Acronym: SGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Michael A. Nielsen, department manager, Copenhagen University Hospital at Herlev
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-D-2008-125
Record Dates: First submitted 2011-03-17; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Malnutrition
Keywords: Nutrition; new energy dense food concept
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nutritional intervention (Experimental)
  Interventions: Dietary Supplement: Nutritional intervention

INTERVENTIONS:
Dietary Supplement: Nutritional intervention — The study was a 12 weeks intervention trial with inclusion of 40 patients at nutritional risk, according to the NRS-2002 system.
  All included patients received nutritional counseling and information about the new food concept by a clinical dietician.
  Recording of the dietary intake was carried out on a daily basis over a period of 3 to 7 days, with nutritional registration forms filled in by the nurse and/or the patient.

SUMMARY:
Rationale:

The objective of this study was to investigate whether a new energy dense food concept, on order 24 hours a day, would lead to a minimum 75% intake of nutritional needs in patients at nutritional risk. The investigators target was for 70% of patients to reach 75% of their energy and protein requirements.

Methods:

An intervention study was conducted with inclusion of 40 patients at nutritional risk, according to the NRS-2002 criteria. The food concept consisted of 36 small delicious dishes. Patients could choose food from both the new concept and the ordinary patient buffet. The investigators monitored patients' nutritional requirements and daily nutritional intake.

ELIGIBILITY:
Inclusion Criteria:

* patients at nutritional risk, according to the NRS-2002 criteria.
* patient must be able to understand the information and be able to give a written inform consent
* well-functioning gastrointestinal tract
* Anticipated length of hospitalization > 5 days
* Should understand and speak danish

Exclusion Criteria:

* Terminal patients
* patients with dysphagia
* patient with food allergy or intolerance
* patients who only receives enteral or parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change in energy and protein intake compared to the historical control group | 3 to 7 days recording of dietary intake
  The patient's energy requirement was estimated both from the factorial method and by Harris and Benedicts formula and the protein requirements was taken to be 18 E % of the energy requirement.
  Recording of the dietary intake was carried out on a daily basis over a period of 3 to 7 days, with nutritional registration forms filled in by the nurse and/or the patient. The nutritional registration forms contained information of the energy and protein content of the food

CONTACTS AND LOCATIONS:
Overall Officials: Tina Munk, MSc., Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen University Hospital at Herlev, Herlev, Denmark